CLINICAL TRIAL: NCT05804955
Title: Alpha-Glutathione-S-Transferase (AlphaGST) and the MARINA Index as a Novel Predictive Biomarker and Composite Tool for Disease Impairment in the MASLD Context
Brief Title: Alpha-Glutathione-S-Transferase (AlphaGST) and MARINA Index in Metabolic-Dysfunction-Associated-Steatotic-Liver-Disease (MASLD)
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Alessandro Federico, Professor, University of Campania Luigi Vanvitelli
Other Study IDs: 530/2016
Record Dates: First submitted 2023-03-03; First posted 2023-04-07 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Fatty Liver
Keywords: Metabolic dysfunction Associated Steatotic Liver Disease; liver fibrosis; liver cirrhosis; non-invasive biomarkers; cardiovascular risk
MeSH Terms: conditions — Fatty Liver; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum and biopsy liver samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training Cohort: 200 MASLD patients
- Validation Cohort: 60 MASLD patients

SUMMARY:
AlphaGST represents a liver enzyme whose serologic levels progressively increase in alcoholic and viral chronic hepatitis according to the worsening of liver fibrosis. However, its diagnostic and prognostic usefulness in Metabolic-dysfunction-Associated-Steatotic-Liver-Disease has never been explored.

The investigators aimed to assess the alphaGST levels in Metabolic-dysfunction-Associated-Steatotic-Liver-Disease patients affected by different stages of liver fibrosis, and, by using a new-designed "Metabolic Abnormalities Related to lipids- Insulin resistance-AlphaGST levels" (MARINA) index, to evaluate its role as a novel non-invasive tool in the disease staging stratification, identification of the advanced fibrosis and prediction of 5-years acute cardiovascular events occurrence.

The investigators enrolled 30 ehalthy controls and 200 metabolic dysfunction-associated steatotic liver disease patients (Training cohort) (TrC). As a validation cohort (VlC), between January 2018 and May 2019, 60 MASLD patients were consecutively enrolled (Validation Cohort - VlC) All Metabolic-dysfunction-Associated- Steatotic-Liver-Disease patients received an ultrasound-guided percutaneous liver biopsy for the disease staging. Liver stiffness measurement, NAFLD fibrosis score, Fibrosis-4, and body mass index-aspartate aminotransferase/Platelet Ratio-Diabetes scores as well as the MARINA index were determined. Naïve-acute cardiovascular events patients were subsequently followed up over 5 years to record acute cardiovascular events occurrence.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years
* MASLD diagnosis

Exclusion Criteria:

* presence of chronic inflammatory diseases
* acute or chronic kidney diseases
* rheumatoid arthritis, systemic lupus erythematosus, or other major systemic inflammatory diseases or tumors
* ongoing infections
* alcohol or drug abuse history
* other etiologies of chronic liver damage
* previous hepatocellular carcinoma diagnosis
* use of hepatoprotective drugs
* decompensated liver cirrhosis (Child-Pugh B and Child-Pugh C) at the moment of the enrollment or in the previous 12 months
* psychological/psychiatric problems that could have invalidated the informed consent

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: After signing the informed consent, the investigators consecutively enrolled patients affected by ultrasonographic detectable bright-liver presenting the MAFLD diagnostic features:1) overweight or obesity, defined as Body Mass Index >25 kg/m2; 2) type 2 diabetes mellitus; 3) presence of ≥ two metabolic risk abnormalities identified by (a) waist circumference ≥102 cm in men (≥ 88 cm in women), (b) blood pressure ≥ 130/85 mmHg (or specific drug treatment), (c) plasma triglycerides ≥150 mg/dL (or specific drug treatment), (d) plasma high-density-lipoprotein cholesterol < 40 mg/dL for men (<50 mg/dL for women) (or specific drug treatment), (e) prediabetes (fasting plasma glucose levels 100-125 mg/dL) or 2-hour post-load glucose levels 140-199 mg/dL or glycated hemoglobin 5.7%-6.4%, (f) homeostasis-model-assessment-for-insulin-resistance score ≥2.5, (g) plasma high-sensitivity C-reactive protein level > 2 mg/L.
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Alpha-Glutathione-S-Transferase (alpha GST) prediction of advanced fibrosis | baseline
  The diagnostic accuracy of the alpha-Glutathione-S-Transferase (alphaGST) blood levels (pg/ml) in the prediction of hepatic histological-proved advanced fibrosis
MARINA Index prediction of advanced fibrosis | baseline
  The diagnostic accuracy of the MARINA index in the prediction of hepatic histological-proved advanced fibrosis. The MARINA index was calculated by combining the following variables: HLD > 43.5 mg/dl (no: 1 point; yes: 2 points); HbA1c > 5.5% (no: 1 point; yes: 2 points); AlphaGST > 3917 pg/ml (no: 2 point; yes: 4 point). MARINA index total scores ranged from 3 to 8 points.

SECONDARY OUTCOMES:
MARINA index in the prediction of acute cardiovascular events | five years
  The accuracy of the MARINA index in the prediction of Acute Cardiovascular Events 5 years occurrence. The MARINA index was calculated by combining the following variables: HLD > 43.5 mg/dl (no: 1 point; yes: 2 points); HbA1c > 5.5% (no: 1 point; yes: 2 points); AlphaGST > 3917 pg/ml (no: 2 point; yes: 4 point). MARINA index total scores ranged from 3 to 8 points.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Federico, Professor, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- University of Campania Luigi Vanvitelli, Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data (IPD) that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: six months after the acceptance for 10 years
Access Criteria: upon reasonable request to the corresponding author